CLINICAL TRIAL: NCT02988934
Title: The WATS3D (Wide Area Transepithelial Sample Biopsy With 3-Dimensional Computer-Assisted Analysis) U.S. Registry
Status: Terminated | Type: Observational
Sponsor: CDx Diagnostics (Industry)
Collaborators: University of North Carolina, Chapel Hill (Other)
Responsible Party: Sponsor
Other Study IDs: CDx 707
Record Dates: First submitted 2016-11-29; First posted 2016-12-12 (Estimated); Last update posted 2023-02-08 (Actual); Status verified 2023-02

CONDITIONS: Barrett Esophagus; Gastroesophageal Reflux; Esophageal Dysplasia; Esophageal Diseases
MeSH Terms: conditions — Barrett Esophagus; Gastroesophageal Reflux; Esophageal Diseases

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 10 Years

SUMMARY:
The purpose of this study is to create a registry (collect data and keep it in a research database) to learn more about two methods of taking small tissue samples from your esophagus (the esophagus is the tube that carries food and liquid from your mouth to your stomach.). The two methods of sampling are: 1) Using forceps that take biopsies (small tissue samples) from your esophagus, and 2) Using a brush that also takes biopsies from your esophagus.

By recording the results of all of your biopsies over many years, it may be possible to find out if the brush biopsy, forceps biopsy, or both can predict which patients with heartburn develop Barrett's esophagus, (an abnormality in the esophagus that may lead to cancer), and which patients with Barrett's esophagus develop precancer and cancer. The data from your biopsies will be used to determine the best way to diagnose esophageal disease.

You are being asked to participate in the study because you are receiving an upper endoscopy (a procedure where a tube with a light and camera are inserted in your mouth and down your throat) with forceps and brush biopsies of your esophagus as part of your standard clinical care, and you are between the ages of 18 and 80.

ELIGIBILITY:
Inclusion Criteria:

* English speaking
* Able to read, comprehend, and complete the consent form
* Aged 18 to 80, and,
* Meet one of the following:
* Patients with heartburn or regurgitation undergoing a screening EGD, who undergo WATS3D sampling and forceps biopsies for suspicion of BE, or
* Patients with known BE with or without dysplasia undergoing a surveillance EGD with WATS3D biopsies and forceps biopsies, or
* Patients who have undergone endoscopic eradication therapy(including, but not limited to endoscopic mucosal resection, endoscopic submucosal dissection, radiofrequency ablation and/orcryoablation/spray cryotherapy)who are undergoing surveillance EGD following the establishment of complete eradication of intestinal metaplasia (CEIM) with accompanying WATS3D sampling and forceps biopsies.

Exclusion Criteria:

* Patients meeting any of the following criteria will be excluded from this study:
* Patients who on their enrollment endoscopy have a visible highly suspicious lesion, such as a nodule or ulcer, (noted while undergoing endoscopy) that requires targeted biopsy will be excluded from the study.Patients requiring a targeted biopsy on follow-up endoscopies will be allowed to remain in the study.
* Patients who do not undergo both biopsy forceps and WATS3D biopsy of the esophagus on their initial evaluationfor routine care will be excluded from this study. Subsequent endoscopicevaluation may include forceps biopsies alone, WATS3D biopsies alone, or both forceps and WATS3D biopsies.

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: males and females
Sampling Method: Probability Sample
Enrollment: 3173 (Actual)
Dates: Start 2016-04; Primary Completion 2023-02-07 (Actual); Study Completion 2023-02-07 (Actual)

PRIMARY OUTCOMES:
Incremental yield for dysplasia due to WATS sampling above that noted from routine forceps biopsies in various clinical settings. | 10 years

SECONDARY OUTCOMES:
Outcomes of patients undergoing WATS sampling. | 10 years

CONTACTS AND LOCATIONS:
Locations (1):
- University of North Carolina at Chapel Hill, Chapel Hill, North Carolina, United States